CLINICAL TRIAL: NCT07249294
Title: Multidisciplinary Program to Avoid NSAIDs or Metamizole (HepatoAINEs Study) in Patients With Advanced Chronic Liver Disease Undergoing Major Surgery
Brief Title: Program to Avoid NSAIDs in Patients With Advanced Chronic Liver Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, José Antonio Carrion, Prof. MD. PhD., Parc de Salut Mar
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HepatoAINEs
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Advanced Chronic Liver Disease; Portal Hypertension Related to Cirrhosis
Keywords: Multidisciplinary; Advanced Chronic Liver Disease; Surgery; NSAIDs; Metamizole

STUDY DESIGN:
Intervention Model Description: Prospective interventional study with single-group assignment. A historical cohort will be used for external comparison but is not part of the randomized arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prevention Strategy (Experimental): Participants with cirrhosis will receive an intervention designed to prevent the administration of non-steroidal anti-inflammatory drugs (NSAIDs), which are contraindicated in this population. The intervention includes clinical alerts, prescriber education, and pharmacy verification steps. Outcomes will be compared to a historical cohort of cirrhotic patients who were exposed to NSAIDs prior to implementation of the preventive strategy.
  Interventions: Behavioral: Multidisciplinary support program

INTERVENTIONS:
Behavioral: Multidisciplinary support program — The intervention includes guideline updates, automated alerts, and multidisciplinary support program (MSP) with collaboration among Digestive, Anesthesia, Surgery, and Pharmacy services to avoid the use of NSAIDs or metamizole in patients with cirrhosis.

SUMMARY:
This study aims to implement measures to avoid the use of NSAIDs or metamizole in patients with advanced chronic liver disease (ACLD) scheduled for major surgery, which are contraindicated due to increased risk of renal dysfunction such as acute kidney injury (AKI), clinical decompensation such as ascites, and bleeding.

DETAILED DESCRIPTION:
The "HepatoAINEs" program introduces information and communication technologies (ICTs) to identify patients with ACLD and prevent NSAIDs/metamizole prescription during perioperative care. The intervention includes guideline updates, automated alerts, and multidisciplinary support program (MSP) with collaboration among Digestive, Anesthesia, Surgery, and Pharmacy services to avoid the use of NSAIDs or metamizole in patients with ACLD scheduled for major surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years) with ACLD scheduled for major surgery
* Exclusion Criteria: Absence of ACLD or portal hypertension, lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
NSAIDs/metamizole prescription | 180 days
  rate of NSAIDs/metamizole prescriptions in patients with ACLD after surgery

SECONDARY OUTCOMES:
complications | 180 days
  rate of AKI, ascites, bleeding, and mortality in patients with ACLD after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Canillas L, Pelegrina A, Alvarez J, Colominas-Gonzalez E, Salar A, Aguilera L, Burdio F, Montes A, Grau S, Grande L, Carrion JA. Clinical Guideline on Perioperative Management of Patients with Advanced Chronic Liver Disease. Life (Basel). 2023 Jan 3;13(1):132. doi: 10.3390/life13010132. PMID 36676081